CLINICAL TRIAL: NCT02743533
Title: Trends in the Incidence, Treatment and Prognosis of Cardiovascular Diseases in the Silesian Region in Poland. SILesIan CARdiovascular Database (SILICARD)
Brief Title: Cardiovascular Diseases in the Silesian Region in Poland.
Acronym: SILICARD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Silesian Centre for Heart Diseases (Other)
Responsible Party: Principal Investigator, Mariusz Gasior, Professor, PhD, Silesian Centre for Heart Diseases
Other Study IDs: SCD016
Record Dates: First submitted 2016-04-04; First posted 2016-04-19 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Cardiovascular Diseases
Keywords: cardiovascular diseases, prognosis
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The Silesian Cardiovascular Database is an observational study of all patients hospitalized due to cardiovascular diseases. The date include information on the clinical characteristics, treatment modalities and prognosis in this population.

The data include information on all the applicable diagnostic and therapeutic procedures, prognosis and hospitalization costs. Likewise, data have been collected specialist care outpatient visits and primary health care patients were hospitalized.

DETAILED DESCRIPTION:
The Silesian Cardiovascular Database is an prospective observational study patients who were hospitalized in the Silesian region in Poland due to cardiovascular diseases from 1st January 2006.

The aim of the study is to collect and analyze all epidemiological data, diagnostic and therapeutic procedures, in-hospital and long-term prognosis, hospitalization costs of these patients. Likewise, data have been collected specialist care outpatient visits and primary health care patients were hospitalized.

For the analysis were included patients hospitalized in the cardiology, cardiac surgery , diabetes, vascular surgery wards and who were hospitalized for cardiac diagnosis in the wards of internal medicine and intensive care.

The Silesian Cardiovascular Database was created based on the agreement between Silesian Centre for Heart Diseases in Zabrze and the Regional Department of National Health Fund in Katowice in order to conduct analyses and prepare scientific elaborations on the group of patients with circulatory system diseases. Data elaboration and preparation for analyses was conducted by the Science Department of Silesian Centre for Heart Diseases and the Department of Biostatistics of Medical University of Silesia.

ELIGIBILITY:
Inclusion Criteria:

* each hospitalisation in the departments of: cardiology, cardiac surgery, diabetology and vascular surgery,
* hospitalisation with cardiological diagnosis in the departments of internal medicine and intensive care.

Exclusion Criteria:

* hospitalisations of patients from beyond Silesia Province,
* patients at the age below18 years at the moment of admission to the hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is formed by all patients hospitalized in the Silesian region in Poland due to cardiovascular diseases from 1st January 2006.
Sampling Method: Non-Probability Sample
Enrollment: 10000000 (Estimated)
Dates: Start 2006-01; Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with reported deaths from any cause | From date of inclusion until the date of death from any cause, assessed up to 1 year

SECONDARY OUTCOMES:
Trends in the number of hospitalization due to cardiovascular diseases | 1 year
Trends in the number of diagnostic and therapeutic procedures | 1 year
Number of participants with reported rehospitalization | From date of inclusion until the date of first event, assessed up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mariusz Gasior, Prof., PhD, Principal Investigator — 3rd Chair and Department of Cardiology, Silesian Center for Heart Diseases, Zabrze, Poland; Damian Pres, MD, Study Chair — 3rd Chair and Department of Cardiology, Silesian Center for Heart Diseases, Zabrze, Poland
Locations (1):
- Silesian Center for Heart Diseases, Zabrze, Poland

REFERENCES:
- [Derived] Myrda K, Blachut A, Buchta P, Skrzypek M, Wnuk-Wojnar AM, Hoffmann A, Nowak S, Kowalski O, Pruszkowska P, Sokal A, Wita K, Mizia-Stec K, Gasior M, Kalarus Z. Impact of the coronavirus disease 2019 pandemic on atrial fibrillation and atrial flutter ablation rates. The analysis of nearly 5 million Polish population. Kardiol Pol. 2021;79(6):687-689. doi: 10.33963/KP.15988. Epub 2021 May 20. No abstract available. PMID 33926171